CLINICAL TRIAL: NCT07398404
Title: A Multiple Health Behavior Change Intervention for Weight Loss and Smoking Cessation for Pre-Bariatric Surgery Patients
Brief Title: A Multiple Health Behavior Change (MHBC) Intervention for Weight Loss and Smoking Cessation for Pre-Bariatric Surgery Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000041823
Record Dates: First submitted 2026-01-28; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Smoking Cessation; Bariatric Surgery Patients
MeSH Terms: conditions — Obesity; Smoking Cessation | interventions — Naltrexone; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the active intervention group or the standard of care control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MHBC Intervention Group (Experimental): Participants will receive the multiple health behavior intervention with combined behavioral and pharmacotherapy (Naltrexone/Bupropion).
  Interventions: Drug: Naltrexone hydrochloride; Drug: Bupropion Hydrochloride Extended-release; Behavioral: Cognitive-Behavioral Therapy
- Control Group (No Intervention): Participants will receive the current standard of care treatments and services offered by the bariatric clinic for weight loss and smoking cessation.

INTERVENTIONS:
Drug: Naltrexone hydrochloride — Participants will be given 50mg/day of Naltrexone for 4 months.
  Arms: MHBC Intervention Group
Drug: Bupropion Hydrochloride Extended-release — Participants will be given 300mg/day of Bupropion for 4 months. Bupropion will be taken twice daily (150mg in the morning, followed by 150mg in the late afternoon/early evening).
  Arms: MHBC Intervention Group
Behavioral: Cognitive-Behavioral Therapy — Participants will receive cognitive-behavioral therapy for weight loss and smoking cessation. Participants will meet with their assigned study clinician weekly for 60 minutes for 4 months.
  Arms: MHBC Intervention Group

SUMMARY:
The purpose of this research study is to evaluate a multiple health behavior change intervention for weight loss and smoking cessation using medication (Naltrexone + Bupropion) and behavior therapy in adults seeking bariatric surgery. The intervention will be compared to a standard of care control group.

DETAILED DESCRIPTION:
Smoking prevalence among pre-bariatric surgery patients is estimated to be as high as 40%. In addition to quitting smoking, patients are expected to lose weight before surgery, which is challenging as smoking cessation is associated with weight gain. This study aims to evaluate a multiple health behavior change intervention with combined behavioral and pharmacotherapy (Naltrexone/Bupropion) for weight loss and smoking cessation for adults seeking bariatric surgery. This pilot randomized control trial will evaluate feasibility and acceptability of the intervention and compare the intervention to a standard of care control group.

ELIGIBILITY:
Inclusion Criteria:

* Be 18-65 years old.
* Be actively considering bariatric surgery.
* Smoke at least 5 cigarettes daily for the past 3 months.
* Have a BMI ≥ 30.0 kg/m2.
* Not currently taking medications that interact with Naltrexone or Bupropion (e.g., opiates, benzodiazepines).
* No history of medical conditions that are contraindicated with Naltrexone or - Bupropion (e.g., seizure disorders, uncontrolled hypertension, cardiac issues including history of heart attacks, heart disease, or stroke, history of anorexia or bulimia nervosa).
* Physically well enough to participate in the intervention (e.g., able to walk independently).
* Speak/read/write in English.
* Not currently pregnant or breastfeeding or have plans to become pregnant or breastfeed during the study.
* No active suicidal or homicidal ideation.

Exclusion Criteria:

* Has an acute medical or psychiatric disorder that would make participation difficult or unsafe.
* Has suicidal or homicidal ideation that requires immediate attention.
* Has a predisposition to seizures (e.g., subject with a history or evidence of seizure disorder, febrile seizures during childhood, brain tumor, cerebrovascular disease, or significant head trauma; has a family history of idiopathic seizure disorder or is currently being treated with medications or treatment regimens that lower seizure threshold).
* Has evidence of a second or third degree heart block, atrial fibrillation, atrial flutter, prolongation of the QTc, or any other finding on the screening electrocardiogram that would preclude safe participation.
* Has stage 2 hypertension (blood pressure greater than 160/100 or heart rate over 100 beats/minute).
* Has elevated bilirubin test or any other liver function test value > 5 times the upper limit of normal laboratory criteria.
* Has a platelet count < 100x10 3/uL.
* Has a history of anorexia nervosa or history of bulimia nervosa.
* Is currently taking a medication that is contraindicated to Naltrexone or Bupropion (e.g., MAOIs, opiates).
* Has a history of allergy or sensitivity to Naltrexone or Bupropion.
* Has a co-existing psychiatric condition that requires hospitalization or more intensive treatment (such as bipolar mood disorders, psychotic illnesses, or severe depression).
* Has a history of congenital heart disease, cardiovascular disease, cardiac arrhythmias requiring medication, or a history of cerebrovascular pathology including stroke.
* Has current uncontrolled Type I or Type 2 diabetes mellitus.
* Has a history of severe renal, hepatic, neurological, chronic pulmonary, or gallbladder disease, or any other unstable medical disorder, including cancer.
* Has angle closure glaucoma.
* Has taken an investigational drug in another study within 30 days of study consent.
* Has been prescribed and taken Naltrexone or Bupropion within 30 days of study consent.
* Is concurrently enrolled in formal behavioral or pharmacological Substance Use Disorder treatment.
* Is receiving ongoing treatment with tricyclic antidepressants, xanthines, systemic corticosteroids, nelfinavir, efavirenz, chlorpromazine, MAOIs, central nervous stimulants, or any medication that could interact adversely with the study medications.
* Has a current pattern of alcohol, benzodiazepine, or other sedative hypnotic use which would preclude safe participation in the study.
* Requires treatment with opioid-containing medications during the study period.
* Has a surgery planned other than bariatric surgery.
* Is currently in jail, prison, or any inpatient overnight facility as required by a court of law or have pending legal action or other legal situation that could prevent participation.
* Is currently pregnant, breastfeeding, or plans to become pregnant during the study, or is not using a reliable form of birth control.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Study enrollment to assess Feasibility | 16 weeks
  Number of participants enrolled out of participants screened.
Mean number treatment sessions attended to assess Feasibility | 16 weeks
  Mean number of treatment sessions attended.
Retention to assess Feasibility | 16 weeks
  Retention will be measured as the percent of participants that attend the post treatment assessment.
Treatment credibility to assess Acceptability | Week 4, Week 8, Week 12, Week 16
  Treatment credibility will be assessed via self-report monthly. Acceptability measured as the percent of participants that agree the intervention is acceptable (0-100%, with higher scores being indicative of higher treatment credibility).
Treatment satisfaction to assess Acceptability | Week 16
  Treatment satisfaction will be assessed via self-report at post-treatment. Acceptability measured as the percent of participants that agree the intervention is satisfactory (0-100%, with higher scores being indicative of higher treatment satisfaction).
Percent weight change | Baseline, Week 16, 6-month follow-up
  Percent weight change will be calculated from baseline to post-treatment, and post-treatment to 6-month follow-up.
Smoking cessation, as measured by exhaled carbon monoxide | Baseline, Week 4, Week 8, Week 12, Week 16, 6-month follow-up
  Smoking cessation will be evaluated biochemically, through mean exhaled carbon monoxide concentration.
Smoking cessation, as measured by timeline followback interview | Baseline, Week 4, Week 8, Week 12, Week 16, 6-month follow-up
  Smoking cessation will be evaluated behaviorally, through point prevalence abstinence data obtained by timeline followback interviews.

SECONDARY OUTCOMES:
Nicotine dependence, as measured by the Fagerstrom Test for Nicotine Dependence | Baseline, Week 16, 6-month follow-up
  The Fagerstrom Test for Nicotine Dependence is a self-report measure that classifies level of nicotine dependence. Participants respond to a series of questions assessing time of first cigarette after waking, difficulty refraining from smoking in places where smoking is prohibited, and frequency of smoking. Total score range 0-10 with higher scores indication more nicotine dependence.
Depressive symptomatology, as measured by the Patient Health Questionnaire-9 | Baseline, Week 16, 6-month follow-up
  The Patient Health Questionnaire-9 is a brief, psychometrically sound, and widely used self-report measure of depression in diverse medical settings. The total score on the PHQ-9 ranges from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
Physical activity, as measured by the Global Physical Activity Questionnaire (GPAQ) | Baseline, Week 16, 6-month follow-up
  GPAQ is a validated self-report assessment of physical activity and sedentary behavior. GPAQ does not have a single fixed total score range but a score is calculated in METs-minutes per day. Participants are classified as "active" if they meet or exceed 600 METs-minutes per week.
Bariatric surgery completion | 6-month follow-up
  Bariatric surgery completion will be assessed at 6-month follow-up, through medical record review.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin E Smith, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow A, Neville A, Kolozsvari N. Smoking in bariatric surgery: a systematic review. Surg Endosc. 2021 Jun;35(6):3047-3066. doi: 10.1007/s00464-020-07669-3. Epub 2020 Jun 10. PMID 32524412